CLINICAL TRIAL: NCT04347798
Title: IMPact of Inflammatory Arthritis on COVID-19 sTudy of the RAPPORT-ONTRAAC and FORCAST Rheumatic Disease Registries
Brief Title: IMPACT: IMPact of Antimalarials on Covid-19 Infections in RAPPORT
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00100000
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-03

CONDITIONS: Covid-19 Infection; Rheumatoid Arthritis; Psoriatic Arthritis; Hydroxychloroquine
Keywords: Rheumatoid arthritis; Psoriatic arthritis; Covid-19; Hydroxychloroquine; Chloroquine; Anti-malarials
MeSH Terms: conditions — COVID-19; Arthritis, Rheumatoid; Arthritis, Psoriatic | interventions — Hydroxychloroquine; Chloroquine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Blood sample for Covid-19 serology, ABO blood type, HLA typing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Inflammatory arthritis patients on biologic + anti-malarial: Patients in northern Alberta receiving hydroxychloroquine or chloroquine +/- other disease modifying anti-rheumatic drug + biologic (anti-TNF inhibitor or anti-IL-6 blocker or B-cell depletor or JAK kinase inhibitor or T-cell c-stimulation inhibitor or IL-17 blocker)
  Interventions: Other: Hydroxychloroquine/Chloroquine
- Inflammatory arthritis patients on biologic + NO anti-malarial: Patients in northern Alberta receiving a biologic (anti-TNF inhibitor or anti-IL-6 blocker or B-cell depletor or JAK kinase inhibitor or T-cell c-stimulation inhibitor or IL-17 blocker) +/- any disease modifying anti-rheumatic drug except for anti-malarials (hydroxychloroquine or chloroquine)

INTERVENTIONS:
Other: Hydroxychloroquine/Chloroquine — Prospective evaluation of development of Covid-19 in inflammatory arthritis patients on biologics with anti-malarials compared to inflammatory arthritis patients on biologics without anti-malarial exposure
  Groups: Inflammatory arthritis patients on biologic + anti-malarial

SUMMARY:
This study aims to evaluate the experience of Alberta patients with inflammatory arthritis who participate in the the RAPPORT-ONTRAAC registry during the COVID-19 pandemic, specifically comparing the experience of those taking anti-malarial medications compared to those who do not. This registry includes approximately 2500 northern Alberta patients with inflammatory arthritis who receive highly complex therapies which may be associated with side effects. This program of data collection and research has been evaluating the effectiveness and safety as well as associated health care costs of rheumatoid and psoriatic arthritis patients since 2004. The principle investigators are based at the University of Alberta while the co-investigators are academic rheumatologists at the University of Alberta. The registry has approximately 900 patients taking anti-malarials combined with their complex therapies and ~ 1500 not on anti-malarials in combination with their complex therapies. We aim to perform a case control study evaluating the impact of anti-malarial drugs (eg. hydroxychloroquine and chloroquine) on the development of COVID-19 compared to those patients who are not on anti-malarial drugs over the next 6-12 months. In addition to frequent e-mail surveys screening for the clinical symptoms of COVID-19 and understanding their concomitant arthritis medication use, we will compare the healthcare outcomes of both groups of arthritis patients with and without COVID-19 for the duration of the pandemic. This information will provide critical information beyond an anecdotal level on whether or not anti-malarials truly provide a protective benefit against COVID-19 or reduce the severity of infection. A blood sample from all participants (Covid-19 positive and negative) will be drawn approximately six months into the study for measurement of antibodies to Covid-19 and possible blood types and HLA alleles. Additionally, this study will be linked to another study "Persistence of SARS-Cov2 in immunocompromised patients" which will specifically evaluate COVID-19 serology and nasopharyngeal swab findings in the subset of patients who develop COVID-19.

DETAILED DESCRIPTION:
PURPOSE:

1. To evaluate the impact of anti-malarial medications (hydroxychloroquine and chloroquine) on the development and severity of COVID-19 infection during the current COVID-19 pandemic in an inception cohort registry of northern Alberta rheumatoid and psoriatic arthritis patients who are on complex biologic therapies for the duration of the pandemic.
2. To further evaluate the impact of all biologic medications currently in the registry on the development and severity of COVID-19 by mechanism of action (eg. TNF antagonism vs IL-6 blockade, etc).

HYPOTHESIS: We hypothesize that the "case" group of patients on concomitant anti-malarial treatment with their biologic agent will have a lower incidence and severity of COVID-19 infection compared to those not on anti-malarials based on anecdotal reports of efficacy of anti-malarials on COVID-19 infection from international reports.

JUSTIFICATION: The COVID-19 pandemic has introduced unforeseen challenges internationally and led to great uncertainty for patients who are immunocompromised, such as patients in the RAPPORT registry. Recent anecdotal reports from other countries have been associated with media and political escalation of the potential benefit of anti-malarial drugs on the course of COVID-19 infection. This has led to threats to the supply of anti-malarials drugs for patients with rheumatic diseases like lupus and rheumatoid and psoriatic arthritis, where the benefits are proven. The RAPPORT inception cohort registry provides a unique opportunity to evaluate the impact of COVID-19 in an immunocompromised population, while also evaluating the potential impact of possible treatments for COVID-19.

OBJECTIVES:

Primary

1. To evaluate the impact of anti-malarial medications (hydroxychloroquine and chloroquine) on the development and severity of COVID-19 infection during the current COVID-19 pandemic in an inception cohort registry of northern Alberta rheumatoid and psoriatic arthritis patients who are on complex biologic therapies for the duration of the pandemic.
2. To further evaluate the impact of all biologic medications currently in the registry on the development and severity of COVID-19 by mechanism of action (eg. TNF antagonism vs IL-6 blockade, etc).

Secondary

1. To evaluate the incidence of COVID-19 versus other infections over the remaining duration of the pandemic in an immunocompromised population.
2. To compare the incidence of COVID-19 versus other infections over the remaining duration of the pandemic in the proportion of patients from the RAPPORT registry who take concomitant anti-malarials versus those patients that do NOT take anti-malarials.
3. To compare the impact of different mechanisms of action of biologic medications within the RAPPORT registry, on the incidence of COVID-19 versus other infections

RESEARCH METHOD/PROCEDURES:

For this case control study, we have identified ~900 patients within the RAPPORT-ONTRAAC registry who are taking concomitant anti-malarial medications with their biologic medication compared to ~ 1500 patients who are NOT taking concomitant anti-malarial medications. The current consent for the RAPPORT-ONTRAAC registry allows patients to be contacted for their potential participation in future studies. Based on this consent, we aim to send a letter to all existing RAPPORT patients inviting them to participate in this study.

This letter will be sent by email to those with an associated email address and by Canada Post mail for those who do not. Similar to previous surveys we have conducted, the letter will provide a synopsis of the current situation with the COVID-19 pandemic and request for the patient to consent to the following: (1) consent to receive email/letters with surveys of their clinical status at week 0 (the first point of contact), week 2, then every 4 weeks until the pandemic is over according to the World Health Organization or most appropriate local declaration and (2) consent to allow the study team access to the patient's medical health records (Connectcare/Netcare) for the duration of the pandemic to provide complete information regarding any healthcare utilization, investigations and outcomes over time. The act of consent will be obtained if the patient answers specifically that the study team can access their records and by the act of completing the survey every time. We will collect a blood sample when the pandemic is over from the consenting patients for consideration of serology testing.

The survey will screen for clinical symptoms of COVID-19 and concomitant status of their inflammatory arthritis and medication use. This information is linked by a unique identifier with the RAPPORT-ONTRAAC registry. The RAPPORT-ONTRAAC registry collects baseline, and at least annual information including patient demographics, ethnicity, disease characteristics, serologies, and patient-reported outcomes evaluating the impact of arthritis on their activities of daily living. With the additional linkage to their electronic medical records, we aim to identify the following: hospitalizations, and laboratory and diagnostic investigations. Access to the entire cohort's electronic medical records will provide the opportunity to capture patients who may not develop any symptoms consistent with COVID and/or may not be keen to participate in ongoing surveys but may be impacted by COVID-19. The subset of patients who develop COVID-19 will be contacted to participate in the associated study (Persistence of SARS-CoV2 in immunocompromised patients; Dr. M. Osman) for more in-depth serological evaluations and nasopharyngeal swabs. At the end of the study, we will collect a blood sample as well to ensure that COVID-19 serological evaluations are completed on asymptomatic individuals who participated in the study.

The survey, developed in collaboration with Infectious Disease experts (Drs. Sonpar, Swartz, Shafran, Singh), will screen for currently recognized signs and symptoms of COVID-19. Additionally, confirmation of current arthritis medication use including all disease modifying anti-rheumatic drugs (DMARDS) as well as biologics will be captured. Surveys will be completed on REDCAP through email link, provided directly on the email or as a hyperlink that the patient can type in if they receive the survey by Canada Post. The REDCAP survey will be developed and housed by EPICORE (Epidemiology and Research Coordinating Center).

For the remainder of the pandemic, electronic medical record and NETCARE searches will be conducted for all consenting patients with pre-specified outcomes and interim investigations and/or procedures or hospitalizations in Alberta Health Services facilities. REDCAP survey responses will be collated with these searches.

PLAN FOR DATA ANALYSIS: A response rate of 40% is expected for this study. Descriptive data analyses will be conducted to describe the population of inflammatory arthritis patients divided between those who are currently taking an anti-malarial and those who are not. The registry provides information including demographics (gender, age, ethnicity) and at least annual disease activity status with validated disease activity scores which differentiate between low disease activity state/remission and mild, moderate and severe disease activity. Co-morbidities through the Charlson Comorbidity Index will be identified and compared between groups. Survey results over the pandemic per patient will be analyzed. Electronic medical records will be reviewed at least monthly for all consenting patients to identify and quantify investigations, procedures and healthcare resources utilized during the pandemic.

With multivariate analyses, the impact of anti-malarial use on the development and severity of COVID-19 will be evaluated between the two groups, adjusting for important confounders including the following: co-morbidities (eg. cardiac and respiratory diseases, diabetes), biologic mediations, steroid use and other DMARDs. Further stratification by biologic DMARD might be conducted. Healthcare utilization between groups will be compared over time. Quantification of antibodies to Covid-19 will be compared between the anti-malarial and non-anti-malarial groups.

ELIGIBILITY:
Inclusion Criteria:

* Current active and consented patient of the Rheumatoid Arthritis Pharmacovigilance Program of Northern Alberta with an e-mail or mailing address

Exclusion Criteria:

* Unable to read English; not consenting to be contacted for future studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult patients with rheumatoid or psoriatic arthritis in northern Alberta who are followed in the RAPPORT registry; all patients are on a biologic agent and possibly one or more disease modifying anti-rheumatic drug (eg. hydroxychloroquine, chloroquine, methotrexate, leflunomide, gold, azathioprine, sulfasalazine)
Sampling Method: Non-Probability Sample
Enrollment: 773 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Impact of anti-malarials on the development and severity of Covid-19 in the anti-malarial group compared to the non-anti-malarial group | 12 months
  Number of patients developing signs and symptoms of Covid-19 or other infections

SECONDARY OUTCOMES:
Incidence of Covid-19 infection in the anti-malarial group compared to the non-anti-malarial group | 12 months
  Number of patients developing Covid-19 infection
Incidence of Covid-19 infection in the sub-groups of patients on biologic agents with different mechanisms of action | 12 months
  Incidence of Covid-19 infection in the sub-groups of patients on biologic agents with different mechanisms of action

OTHER OUTCOMES:
Quantification of Covid-19 antibodies in anti-malarial vs non-anti-malarial groups of inflammatory arthritis patients | 6 months
  Quantitative measurement of Covid-19 serology to understand possible differences in degree of immune response adjusted for anti-malarial and/or biologic exposure

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie O Keeling, MD, Principal Investigator — University of Alberta; Walter P Maksymowych, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada